CLINICAL TRIAL: NCT02418533
Title: A Prospective, Randomized Trial to Compare Mono-menotropins Protocol for Controlled Ovarian Stimulation (COS) Versus Recombinant Follicle Stimulating Hormone (rFSH) Protocol on Embryo Quality Parameters in IVF Patients
Brief Title: Mono-menotropins Versus rFSH Protocol on Embryo Quality
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Main Line Fertility Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MLFC-004
Record Dates: First submitted 2015-03-31; First posted 2015-04-16 (Estimated); Last update posted 2020-08-12 (Actual); Status verified 2020-08

CONDITIONS: Infertility; Fertility
Keywords: infertility; in vitro fertilization; fertility; preimplantation genetic screening; embryo; PGS; Eeva; IVF
MeSH Terms: conditions — Infertility | interventions — Menotropins; follitropin alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mono-menotropin protocol (Experimental): Stimulation Group 1: Mono-Menotropin Protocol Fifty patients will undergo the standard of care COS for IVF using Menopur only. Patients will receive 300 IU of Menopur injected subcutaneously daily for the first five days of stimulation. Thereafter, Menopur may be adjusted (to optimize ovarian response by patient's physician) in 75 IU increments up to a total of 450 IU Menopur daily up to and including day of hCG trigger.
  Interventions: Drug: menotropin
- rFSH protocol (Experimental): Stimulation Group 2: Recombinant follicle stimulating hormone (rFSH) Protocol Fifty patients will undergo the standard of care COS for IVF using Gonal-f (EMD Serono, USA) Protocol. Patients will receive Gonal-f (300 IU) administered subcutaneously daily for the first five days of stimulation. Thereafter, Gonal-f may be adjusted (to optimize ovarian response by the patient's physician) in 75 IU increments up to a total of 450 IU daily up to and including day of hCG trigger.
  Interventions: Drug: Recominant Follicle Stimulating Hormone (rFSH)

INTERVENTIONS:
Drug: menotropin — Menopur is used for controlled ovarian stimulation (COH)
  Other Names: Menopur
  Arms: Mono-menotropin protocol
Drug: Recominant Follicle Stimulating Hormone (rFSH) — Gonal-f is used for controlled ovarian stimulation (COH)
  Other Names: Gonal-f
  Arms: rFSH protocol

SUMMARY:
This study is for couples pursuing in vitro fertilization (IVF) with preimplantation genetic screening (PGS) of embryos to achieve pregnancy. The objective of this clinical trial is to study the effect of mono-menotropins for COS versus recombinant follicle stimulating hormone (rFSH) on cleavage-stage and blastocyst embryo quality after IVF. Embryo quality parameters include conventional embryo grade, early embryo viability assessment (Eeva) time-lapse parameters, and chromosomal aneuploidy rates after PGS.

This pilot study is expected to significantly contribute to optimization of treatment regimens and stimulation protocols to optimize embryo quality.

DETAILED DESCRIPTION:
This proposed study is a single-center, prospective, randomized experimental design.

One-hundred women between the ages of 21 to 38 (inclusive) pursuing IVF treatment for infertility and preimplantation genetic screening (PGS).

Pre-medication All study patients will take oral contraception pills (OCP) starting between day 2-4 of the menstrual cycle before controlled ovarian stimulation (COS) is started for IVF, and they are continued for 21 days. Cycle preparation using an oral contraceptive pill is thought to be important in improving follicular homogeneity.

Randomization Randomization of patients into the Stimulation Group 1 (Mono-Menotropin Protocol) or Stimulation Group 2 (rFSH) will occur at OCP start using a computerized randomization program.

Ovarian Stimulation Stimulation Group 1: Mono-Menotropin Protocol Fifty patients will undergo the standard of care COS for IVF using Menopur (Ferring, Parsippany, New Jersey (NJ) USA) only. Patients will receive 300 IU of Menopur injected subcutaneously daily for the first five days of stimulation. Thereafter, Menopur may be adjusted (to optimize ovarian response by patient's physician) in 75 IU increments up to a total of 450 IU Menopur daily up to and including day of hCG trigger.

Stimulation Group 2: rFSH Protocol Fifty patients will undergo the standard of care controlled ovarian stimulation (COS) for IVF using Gonal-f (EMD Serono, USA) protocol. Patients will receive 300 IU of Gonal-f administered subcutaneously daily for the first five days of stimulation. Thereafter, Gonal-f may be adjusted (to optimize ovarian response by the patient's physician) in 75 IU increments up to a total of 450 IU daily up to and including day of hCG trigger.

Menopur and Gonal-f are widely used in controlled ovarian stimulation cycles for the development of multiple follicles in assisted reproductive technology (ART) programs.

Luteinizing Hormone (LH)-surge Suppression Gonadotropin Releasing Hormone (GnRH) antagonist will be used to suppress endogenous pituitary LH for the prevention of premature LH surges. Patients will receive 0.25 mg/day of Ganirelix Acetate or Cetroelix Acetate when follicle size reaches 12 mm and will continue up to and including day of hCG trigger.

HCG Trigger Human chorionic gonadotropin (hCG) will be used intramuscularly (IM) in both stimulation groups to induce oocyte maturation 36 hours prior to the oocyte retrieval procedure

Cycle Monitoring Cycles will be monitored with follicular ultrasound measurements and serum estradiol concentrations throughout ovarian stimulation. HCG will be given IM when at least three follicles reach a diameter of ≥17 mm. Egg retrieval will be conducted by transvaginal ultrasound 36 h after hCG administration.

Insemination All mature oocytes will have intracytoplasmic sperm injection (ICSI) or standard insemination to achieve fertilization.

Embryo Development Two-pronuclei (2pn) embryos will be placed in the Eeva dish after fertilization check at 16-18 hours post ICSI. To maintain a continuous and uninterrupted imaging process from day 1 through day 3, no media changes or dish removal from the incubator will be permitted. On day 3, imaging will be stopped just before routine embryo grading will be performed according to Society for Assisted Reproductive Technology (SART) standards. Cell number and quality score based on symmetry of cells and percent fragmentation will be recorded. Embryos will be tracked individually. Software will automatically measures cell division timings and provide quantitative information regarding embryo development. Embryo grading day 5 will be performed according to standard operating procedure. Blastocysts will be biopsied on day 5 or 6. Biopsies will be sent to a genetics laboratory (Reprogenetics, New Jersey) for aCGH euploidy testing. Biopsied blastocysts will be vitrified for future frozen embryo transfer (FET) cycle/s, in which euploid blastocyst/s with the correct number of chromosomes will be thawed and transferred back to the uterus in an attempt to achieve pregnancy.

Abnormal embryos (aneuploidy embryos with the incorrect number of chromosomes) may be donated to research or discarded.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing IVF in an attempt to achieve pregnancy.
* Day 2-4 Follicle Stimulating Hormone (FSH) < 10 IU/ml, LH< 12 IU/ml, and estradiol <50 pg/ml on day 2-4 of menstrual cycle
* Antimullerian Hormone > 1.5
* Between 10 and 20 basal antral follicles on day 2-4 of the menstrual cycle
* Body weight >50 kg, with BMI > 18 and < 32 kg/m2

Exclusion Criteria:

* Smokers
* Polycystic ovarian disease
* Endometriosis greater than Stage I
* Testicular aspirated sperm
* Preimplantation Genetic Diagnosis (PGD) for single gene disorder
* Preimplantation Genetic Screening (PGS) banking cycles
* Donor Egg Cycles

Ages: 21 Years to 38 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 109 (Actual)
Dates: Start 2015-03; Primary Completion 2017-04 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Embryo Quality | Embryo quality will be assessed on day 3, 5 and 6 of culture
  Embryo quality parameters include conventional embryo grade, early embryo viability assessment (Eeva) time-lapse parameters, and chromosomal aneuploidy rates after PGS.

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Glassner, MD, Principal Investigator — Main Line Fertility; Sharon H Anderson, PhD, Study Director — Main Line Fertility
Locations (1):
- Main Line Fertility Center, Bryn Mawr, Pennsylvania, United States

REFERENCES:
- See also: Main Line Fertility website — http://mainlinefertility.com